CLINICAL TRIAL: NCT07115277
Title: A Single-arm, Multicenter, Phase III Clinical Trial , Evaluate the Diagnostic Performance and Safety of Flotufolastat F-18 Injection PET Imaging in Prostate Cancer Subjects With Biochemical Recurrence Following Prior Treatment
Brief Title: Diagnostic Efficacy and Safety of Flotufolastat F-18 Injection in Subjects With Biochemical Recurrence of Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XTR020-301
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All prostate cancer subjects will undergo PET imaging using Flotufolastat F-18 Injection (Experimental)
  Interventions: Drug: Flotufolastat F-18 Injection

INTERVENTIONS:
Drug: Flotufolastat F-18 Injection — All patients will receive one injection of Flotufolastat F-18 Injection, a PET radiopharmaceutical selective for PSMA. For the injection, subjects will receive a target dose of 8 mCi (296 MBq) ± 20% IV as a bolus injection. Flotufolastat F-18 Injection will be followed by a 10 ml saline flush.

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic performance and safety of Flotufolastat F-18 injection PET imaging in prostate cancer subjects with biochemical recurrence following prior treatment. The main question it aims to answer is:

• What is the correct detection rate of Flotufolastat F 18 injection PET visual reading results compared to the truth standard?

Participants will:

* Receive Flotufolastat F-18 injection
* Undergo PET/CT scanning

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form. 2. Male, aged ≥18 years. 3. Has previously received one or more of the following treatments:

1. Radical prostatectomy (RP);
2. RP with adjuvant radiotherapy (RT);
3. RP with adjuvant androgen deprivation therapy (ADT);
4. Radical RT or focal gland therapy (e.g., brachytherapy, high-intensity focused ultrasound [HIFU]).

   4. Clinically suspected BCR, serum PSA levels should meet at least one of the followings:
   1. After RP with or without adjuvant or salvage therapy: PSA≥ 0.2 ng/mL, and subsequent confirmation that PSA ≥ 0.2 ng/mL.
   2. After RT as primary treatment: PSA increased at least 2 ng/mL compaire to the nadir.
   3. After focal gland therapy as primary treatment: PSA increased at least 2 ng/mL compaire to the nadir.

   5. If positive lesions are detected on the XTR020 PET imaging or conventional imaging, the subject is willing to receive histopathological confirmation or the sequqnce of conventional imaging confirmation.

   6. Male subjects with reproductive potential must use effective contraception during the study period and 6 months after the study completed; their partners should agree to use contraception during the study period and 6 months after the study completed , too.

   Exclusion Criteria:
   1. Planned to receive an X-ray contrast agent or other radioactive imaging agent within 24 hours before XTR020 PET imaging.
   2. Participation in an interventional clinical trial involving a new drug or treatment within 30 days or 5 biological half-lives of the drug prior to XTR020 PET imaging (whichever is longer).
   3. Known allergy to the active ingredient or any excipient of XTR020.
   4. Claustrophobia or inability to tolerate imaging examinations for any other reason.
   5. Poor compliance or deemed unsuitable for participation in this study by the investigator.
   6. Any condition that, in the opinion of the investigator, may interfere with data collection or prevent the study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of Flotufolastat F-18 Injection PET imaging in Chinese prostate cancer subjects with biochemical recurrence (BCR) | 90 days
  Correct Detection Rate (CDR) at the individual level of Flotufolastat F-18 Injection PET imaging in prostate cancer subjects with BCR

SECONDARY OUTCOMES:
To evaluate other diagnostic performance parameters of Flotufolastat F-18 Injection PET imaging in Chinese prostate cancer subjects with BCR | 90 days
  Positive predictive value (PPV) of Flotufolastat F-18 Injection PET imaging at the individual level in prostate cancer subjects with BCR.
  PPV and CDR of Flotufolastat F-18 Injection PET imaging in the prostate bed, pelvic lymph nodes, and three other regions in Chinese prostate cancer subjects with BCR.
To evaluate the diagnostic performance of Flotufolastat F-18 Injection PET imaging in different subgroups of Chinese prostate cancer subjects with BCR | 90 days
  Individual-level PPV and CDR of Flotufolastat F-18 Injection PET imaging in subjects whose baseline conventional imaging is negative.
  Individual-level PPV and CDR of Flotufolastat F-18 Injection PET imaging at different PSA levels.
To evaluate inter-reader and intra-reader interpretative consistency among independent blinded readers. | 90 days
  Kappa values for inter-reader and intra-reader agreement in the interpretation of the same Flotufolastat F-18 Injection PET imaging by different independent blinded readers and by the same reader at different times.
To evaluate the safety of Flotufolastat F-18 Injection . | 3 days
  The types, severity, frequency, and outcomes of adverse events/serious adverse events reported during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No